CLINICAL TRIAL: NCT04612335
Title: Device-based Rate Versus Rhythm Control Treatment in Patients With Symptomatic Recent-onset Atrial Fibrillation in the Emergency Department (RACE 9 OBSERVE-AF)
Brief Title: Device-based Rate Versus Rhythm Control in Symptomatic Recent-onset Atrial Fibrillation (RACE 9 OBSERVE-AF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Dutch Heart Foundation (Other); Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL73104.068.20
Record Dates: First submitted 2020-08-17; First posted 2020-11-02 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Cardiac arrhythmia; Cardioversion; Electrical cardioversion; Watchful waiting; Wait-and-see; Telemonitoring
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Heart Rate; Electric Countershock

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Watchful waiting (Experimental): the watchful-waiting approach consists of administration of rate control medication to obtain relief of symptoms and a heart rate <110 beats per minute, followed by a telemetric rhythm monitoring period of four weeks to guide rate control therapy.
  Interventions: Other: Rate control
- Routine care (Other): Routine care consists of the standard treatment for an acute episode of recent-onset symptomatic atrial fibrillation, namely acute or delayed cardioversion, followed by a telemetric rhythm monitoring period of four weeks to guide rate control therapy.
  Interventions: Other: Pharmacological or electrical cardioversion

INTERVENTIONS:
Other: Rate control — Rate control drugs are administered to obtain symptom relief and a heart rate of <110 bpm, followed by a 4-week telemonitoring period.
  Arms: Watchful waiting
Other: Pharmacological or electrical cardioversion — Pharmacological or electrical cardioversion is performed to achieve restoration of sinus rhythm, either acutely or in a wait-and-see approach, all within 48 hours, and followed by a 4-week telemonitoring period.
  Arms: Routine care

SUMMARY:
Continuous heart rhythm monitoring elucidated the recurrent and transient nature of recent-onset atrial fibrillation (AF). The RACE7 ACWAS showed that a wait-and-see approach (WAS) in patients with recent-onset AF (rate control for symptom relief followed by delayed cardioversion if needed <48h) allows spontaneous conversion to sinus rhythm in 69% of patients, obviating active cardioversion. Recurrences within one month were seen in 30% of patients in both groups, i.e. the initially chosen strategy did not affect the recurrence pattern. Considering the latter, it remains unclear whether cardioversion is needed at all, especially since cardioversion strategy does not seem to affect behaviour of the arrhythmia over time. Instead of cardioversion a watchful-waiting rate control strategy may be appropriate as initial strategy. This allows observing the electrical and clinical behavior of arrhythmia, providing a solid basis for comprehensive and effective early rhythm control. This study is a multi-center clinical randomized controlled trial to show non-inferiority of watchful-waiting with rate control versus routine care in terms of prevalence of sinus rhythm at 4 weeks follow-up, using a novel telemonitoring infrastructure to guide rate control during follow-up.

DETAILED DESCRIPTION:
Until recently standard of care for patients with recent-onset atrial fibrillation (AF) was early cardioversion. This has just been expanded with a delayed cardioversion approach. However, considering the recurrent and transient nature of AF, cardioversion might not be needed at all and rate control medication might be sufficient to accomplish spontaneous conversion to sinus rhythm. The aim of this trial is to evaluate effectiveness (presence of sinus rhythm) of a watchful-waiting approach, i.e. symptom reduction through rate-control medication and monitoring until spontaneous conversion is achieved compared to routine care, consisting of either early or delayed cardioversion. The trial is a multicentre prospective, randomized, open label, non-inferiority trial comparing the interventional watchful-waiting approach to routine care (control).The primary endpoint (presence of sinus rhythm), will be assessed after 4 weeks. The total follow-up time is 1 year.

ELIGIBILITY:
Inclusion Criteria:

* ECG with atrial fibrillation
* Duration of the current AF episode <36 hours
* Symptoms due to atrial fibrillation
* Age > 18 years
* Able and willing to sign informed consent
* Able and willing to use telemetric rhythm recorder

Exclusion Criteria:

* History of persistent AF (episode of AF lasting more than 48 hours and terminated by cardioversion)
* Deemed unsuitable for participation by attending physician
* Hemodynamic instability (heart rate >170 bpm, systolic blood pressure <100 mmHg)
* Acute heart failure
* Signs of myocardial infarction
* History of syncope of unexplained origin
* History of untreated Sick Sinus Syndrome
* History of untreated Wolff-Parkinson-White syndrome
* Currently enrolled in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Presence of sinus rhythm | 4 weeks after inclusion
  Sinus rhythm documented on a 12-lead ECG

SECONDARY OUTCOMES:
Implementation of the telemonitoring infrastructure | 4 weeks
  e.g. use of telemonitoring infrastructure during the 4 weeks follow up, accuracy of alert system
MACCE: major cardiovascular mortality and cardiovascular and cerebrovascular events | 1 year
  e.g. hospitalisation for stroke, myocardial infarction
AF recurrences/AF progression | 4 weeks and 1 year
  e.g. number of AF recurrences, progression to persistent AF
Cost-effectiveness | 1 year
  The costs and cost-effectiveness of the new approach will be determined and compared to the costs and cost-effectiveness of routine care.
Questionnaires on quality of life (SF-36) | 1 year
  Questionnaires on quality of life (e.g. SF-36), will be used to assess whether there are differences between the two arms. The SF-36 will be evaluated according to recommendations; scores will be recoded on a scale of 0-100 and averaged. Higher scores indicate better quality of life.
Patient reported experiences | 1 year
  A questionnaire on patient reported experiences with the telemonitoring device will be used to assess whether there are differences between the two arms. There will be both positively orientated, and negatively orientated questionnes which have to be rated on a scale of 1-5.
Rate and rhythm control interventions (number of) | 4 weeks
  Alert- and patient-triggered
Rhythm control interventions | 1 year
  Number of participants with cardioversion, catheter ablation

CONTACTS AND LOCATIONS:
Overall Officials: Harry JG Crijns, MD, PhD, Study Chair — Head of cardiology department, Maastricht University Medical Center; Dominik Linz, MD, PhD, Principal Investigator — Head of cardiac electrophysiology, Maastricht University Medical Center
Locations (14):
- Netherlands (14):
  - Maastricht University Medical Center, Maastricht, Limburg
  - Noordwest Ziekenhuisgroep, Alkmaar, North Holland
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Rijnstate, Arnhem
  - Medisch Spectrum Twente, Enschede
  - Martini Ziekenhuis, Groningen
  - Universitair Medisch Centrum Groningen, Groningen
  - Zuyderland Medisch Centrum, Heerlen
  - Alrijne Ziekenhuis, Leiderdorp
  - St Antonius Ziekenhuis, Nieuwegein
  - Radboud UMC, Nijmegen
  - Antonius Ziekenhuis, Sneek
  - St. Elisabeth TweeSteden Ziekenhuis, Tilburg
  - VieCuri Medical Centre, Venlo

IPD SHARING:
Plan to Share IPD: Yes
All elements from the CRF matching a future project's CRF may be provided for an aggregated analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Well after publication of main paper
Access Criteria: Please contact principal investigator or study chair.